CLINICAL TRIAL: NCT01807169
Title: Recto Colonic Endoscopic Mucosal Resection and Polypectomy Under Clopidogrel: the "MEDOC"Study.
Brief Title: Recto Colonic Endoscopic Mucosal Resection and Polypectomy Under Clopidogrel
Acronym: MEDOC
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 12-AOI-05; 2012-005365-12 (EudraCT Number)
Record Dates: First submitted 2013-03-04; First posted 2013-03-08 (Estimated); Last update posted 2018-08-06 (Actual); Status verified 2018-08

CONDITIONS: Polyps
Keywords: colon; endoscopy; resection; clopidogrel
MeSH Terms: conditions — Polyps | interventions — Endoscopic Mucosal Resection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Colonic polypectomy or endoscopic mucosal resection (Experimental): Resection of colonic polyps using polypectomy tehnique (with electrocoagulation) or mucosal resection (EMR or mucosectomy) with injection of physiological serum thus resection with electrocoagulation
  Interventions: Procedure: Colonic polypectomy or endoscopic mucosal resection (EMR).

INTERVENTIONS:
Procedure: Colonic polypectomy or endoscopic mucosal resection (EMR). — Resection of colonic polyps using polypectomy tehnique (with electrocoagulation) or mucosal resection (EMR or mucosectomy) with injection of physiological serum thus resection with electrocoagulation

SUMMARY:
The endoscopic management of patients on anti platelet agents (APA) is a wide problem, with prevalence of patients on this type of therapy steadily increasing. The benefit / risk balance to stop or continue the APA for the digestive endoscopic procedure confronts us every day in clinical practice to another: the relationship thrombosis / hemorrhage.

Molecules most commonly used today are aspirin and clopidogrel. Current recommendations from the European Society of Gastrointestinal Endoscopy (ESGE) allow the maintenance of aspirin for the polypectomy. Some preliminary data show that the risk of bleeding during endoscopic mucosal resection (EMR) with aspirin is not significantly higher than polypectomy. The concept of polypectomy / EMR without stopping aspirin is progressively accepted and returned gradually to the usual practice. However, these procedures are still not allowed under clopidogrel, or in a dual APA therapy, in the absence of relevant data on the subject in the literature.

It is necessary to achieve a large national multicenter study, to clarify the risk of post recto colonic EMR and polypectomy bleeding in patients under clopidogrel alone or in combination (aspirin and clopidogrel) taking into account the endoscopic preventive measures used in daily practice by endoscopists in expert centers (clip, ligature and loop devices, preventive adrenalin injection).

The aim of the "MEDOC" study is to determine the incidence of immediate and delayed bleeding after colonic polypectomy and / or EMR for patients on clopidogrel.

It is expected in this work an incidence of post-polypectomy bleeding close to that observed during the implementation of these actions in the population without any anti platelet agents.

DETAILED DESCRIPTION:
The endoscopic management of patients on anti platelet agents (APA) is a wide problem, due to the dramatically increasing prevalence of patients on these therapies. The benefit / risk balance to stop or continue the APA for the digestive endoscopic procedure confronts us every day in clinical practice to another: the relationship thrombosis / hemorrhage. The maintenance of an APA is particularly essential for acute coronary episode, but in the long term, in prevention of recurrent thrombotic cardiovascular disease. Molecules most commonly used today are aspirin and clopidogrel.

Current recommendations from the European Society of Gastrointestinal Endoscopy (ESGE) allow the maintenance of aspirin for the polypectomy. Some preliminary data show that the risk of bleeding during endoscopic mucosal resection (EMR) with aspirin is not significantly higher than polypectomy. The concept of polypectomy / EMR without stopping aspirin is progressively accepted and returned gradually to the usual practice. However, these procedures are still not allowed under clopidogrel, or in a dual APA therapy, in the absence of relevant data on the subject in the literature.

However recent studies disrupt this problem for different reasons: i) endoscopic haemostatic preventive measures have demonstrated efficacy in reducing the rate of immediate and delayed bleeding post polypectomy or EMR; ii) the inadequate modification or untimely stopping APA treatment is always complicated by severe vascular thrombosis events in 5% of patients; iii) three retrospective studies relativize the risk of bleeding after a colonic polypectomy under clopidogrel. It is therefore essential to carry out a prospective, large-scale, multicenter, study to clarify the risk of post colonic EMR/polypectomy bleeding in patients under clopidogrel alone or in combination (aspirin and clopidogrel) taking into account the endoscopic preventive measures used in daily practice by endoscopists in expert centers (clip, ligature and loop devices, preventive adrenalin injection).

The aim of the "MEDOC" study is to determine the incidence of immediate and delayed bleeding after colonic polypectomy and / or EMR for patients on clopidogrel.

The study presents an interventional prospective multicentric and national design.

300 patients will be included. The duration of the study inclusions will be 18 months.

It is expected in this work an incidence of post-polypectomy bleeding close to that observed during the implementation of these actions in the population without any anti platelet agents.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years, male or female
* Polypectomy AND / OR mucosectomy (EMR) performed on clopidogrel and/or aspirin during a colonoscopy with inability to defer action
* Taking a single daily dose of clopidogrel long-term (more than 3 months) or under treatment with clopidogrel and aspirin (aspirin < 375 mg more than 3 months) in the prevention of cardiovascular and thromboembolic risk with a major or medium - secondary prevention
* Affiliation to the regime of national health protection
* Informed consent and patient's written obtained
* No participation in another clinical study

Exclusion Criteria:

* Contraindications to the achievement of a lower gastrointestinal endoscopy
* Taking a single daily dose of clopidogrel or other anti-platelet, anti vitamin K (AVK), heparin or anti bi aggregation in the context of cardiovascular prevention
* Taking chronic anti inflammatory drug (at least once weekly)
* Resection technique submucosal dissection
* Haemorrhagic disease, disorders of hemostasis and coagulation (PT <60%, aPTT> 40 sec. And platelets <100000/mm3), hematologic malignancy, chronic liver cirrhosis classified as Child Pugh B or C, acute or chronic renal failure
* Acute Coronary Syndrome <3 months or not received percutaneous coronary intervention (PCI).
* Angioplasty with placement of a stent drug evaluation (out of context of acute coronary syndrome) <3 months.
* Angioplasty with placement of a bare metal stent (out of context of acute coronary syndrome) <4 weeks.
* Pregnant women, nursing
* Not signing the written consent and / or mental disabilities of the subject making its participation in the trial impossible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2013-05-14 (Actual); Primary Completion 2017-11-07 (Actual); Study Completion 2017-11-07 (Actual)

PRIMARY OUTCOMES:
Incidence of delayed bleeding after polypectomy and / or colonic mucosectomy | during surgery, hospitalization and at 30 days
  Incidence of delayed bleeding after polypectomy and / or colonic mucosectomy (endoscopic mucosal resection) in patients on clopidogrel

SECONDARY OUTCOMES:
Incidence of immediate bleeding after polypectomy and / or colonic mucosectomy | during surgery, hospitalization and at 30 days
Incidence of severe bleeding after polypectomy and / or colonic mucosectomy in patients on Clopidogrel | during surgery, hospitalization and at 30 days
Efficacy of endoscopic hemostasis in case of bleeding induced | in case of bleeding induced
  Defined by the cessation of bleeding without the need for further treatment (surgery, radiation)
morbidity / mortality induced by immediate and delayed bleeding after polypectomy and / or colonic mucosectomy in patients on clopidogrel | during surgery, hospitalization and at 30 days
predictors of gastrointestinal bleeding post polypectomy / mucosectomy under clopidogrel by sub groups of patients obtained | during surgery, hospitalization and at 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Geoffroy VANBIERVLIET, MD, Study Director — Centre Hospitalier Universitaire de Nice
Locations (3):
- France (3):
  - Centre Hospitalier Universitaire de Bordeaux, Bordeaux
  - Centre Hospitalier Universitaire de Brest, Brest
  - Centre Hospitalier Universitaire de Nice, Nice